CLINICAL TRIAL: NCT05961657
Title: Hemodynamic Evaluation in Preterm Babies Using UltraSonic Cardiac Output Monitor (USCOM)
Brief Title: USCOM Parameters in Preterm Infants: Reference Ranges
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Responsible Party: Principal Investigator, Daniela Doni, Consultant Neonatologist, Fondazione IRCCS San Gerardo dei Tintori
Other Study IDs: EmoNeo
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Very Low Birth Weight Infant; Very Preterm Maturity of Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hemodynamic measurements by USCOM — We will measure cardiac output, cardiac index, and systemic vascular resistance index on 3, 7, and 14 postnatal days using the UltraSonic Cardiac Output Monitor.

SUMMARY:
The goal of this observational study is to learn about the feasibility of hemodynamic measurement by the UltraSonic Cardiac Output Monitor (USCOM) in very preterm or very-low-birth-weight infants. The main questions it aims to answer are: 1) establishing reference ranges for USCOM parameters in this specific population, 2) assessing the effect of patients' characteristics and other possible confounders on USCOM parameters, and 3) evaluating the short-term repeatability of the measurement. Participants will receive USCOM measurements on 3, 7, and 14 postnatal days.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth below 32 weeks and/or
* birth weight (BW) below 1500 g

Exclusion Criteria:

* congenital heart diseases,
* hemodynamic instability requiring drugs that affect hemodynamics (e.g., inotropes)

Ages: 2 Days to 16 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We include very preterm and/or very low birth weight infants without heart disease as assessed by echocardiography, who are considered hemodynamically stable by the attending physician and do not require drugs that might affect the cardiocirculatory function (e.g., inotropes).
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-08-09 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output at 3 days | 3 ± 1 days of life
  Cardiac Output measured by the USCOM system, normalized by body weight and expressed in ml/kg/min
Cardiac Output at 7 days | 7 ± 2 days of life
  Cardiac Output measured by the USCOM system, normalized by body weight and expressed in ml/kg/min
Cardiac Output at 14 days | 14 ± 2 days of life
  Cardiac Output measured by the USCOM system, normalized by body weight and expressed in ml/kg/min
Cardiac Index at 3 days | 3 ± 1 days of life
  Cardiac Output measured by the USCOM system normalized by body surface and expressed in L/min/m2
Cardiac Index at 7 days | 7 ± 2 days of life
  Cardiac Output measured by the USCOM system normalized by body surface and expressed in L/min/m2
Cardiac Index at 14 days | 14 ± 2 days of life
  Cardiac Output measured by the USCOM system normalized by body surface and expressed in L/min/m2
Systemic Vascular Resistance Index at 3 days | 3 ± 1 days of life
  Systemic Vascular Resistance measured by the USCOM system normalized by body surface and expressed in d*s*cm-5/m2
Systemic Vascular Resistance Index at 7 days | 7 ± 2 days of life
  Systemic Vascular Resistance measured by the USCOM system normalized by body surface and expressed in d*s*cm-5/m2
Systemic Vascular Resistance Index at 14 days | 14 ± 2 days of life
  Systemic Vascular Resistance measured by the USCOM system normalized by body surface and expressed in d*s*cm-5/m2

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Doni, MD, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doni D, Nucera S, Rigotti C, Arosio E, Cavalleri V, Ronconi M, Ventura ML, Fedeli T. Evaluation of hemodynamics in healthy term neonates using ultrasonic cardiac output monitor. Ital J Pediatr. 2020 Aug 5;46(1):112. doi: 10.1186/s13052-020-00872-x. PMID 32758264
- [Background] Patel N, Dodsworth M, Mills JF. Cardiac output measurement in newborn infants using the ultrasonic cardiac output monitor: an assessment of agreement with conventional echocardiography, repeatability and new user experience. Arch Dis Child Fetal Neonatal Ed. 2011 May;96(3):F206-11. doi: 10.1136/adc.2009.170704. Epub 2010 Jul 6. PMID 20605971
- [Background] Fraga MV, Dysart KC, Rintoul N, Chaudhary AS, Ratcliffe SJ, Fedec A, Kren S, Cohen MS, Kirpalani H. Cardiac Output Measurement Using the Ultrasonic Cardiac Output Monitor: A Validation Study in Newborn Infants. Neonatology. 2019;116(3):260-268. doi: 10.1159/000501005. Epub 2019 Jul 19. PMID 31326967
- [Background] He SR, Zhang C, Liu YM, Sun YX, Zhuang J, Chen JM, Madigan VM, Smith BE, Sun X. Accuracy of the ultrasonic cardiac output monitor in healthy term neonates during postnatal circulatory adaptation. Chin Med J (Engl). 2011 Aug;124(15):2284-9. PMID 21933558